CLINICAL TRIAL: NCT00067574
Title: Structured Treatment Interruption as an Autovaccination Approach to Enhance Immune Based HIV-1 Control in an Adolescent/Young Adult Population
Brief Title: Treatment Plan to Decrease Drug Exposure in HIV Infected Adolescents
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was never opened for enrollment; concept became irrelevant as other study results became available.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATN 008
Record Dates: First submitted 2003-08-25; First posted 2003-08-26 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2016-07

CONDITIONS: HIV Infections
Keywords: Structured treatment interruption; Treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Treatment Interruption

INTERVENTIONS:
Behavioral: Structured treatment interruption

SUMMARY:
This study will attempt to stimulate the immune system in HIV infected adolescents and young adults so that it can better control the HIV infection. When anti-HIV drugs are stopped for a period of time, the virus "grows back." This may stimulate the immune system, which may then be more effective in controlling the virus.

DETAILED DESCRIPTION:
The focus of this study is to use Structured Treatment Interruption (STI) as an approach to auto-immunization. The STI management schema is based on current understanding of HIV-1 viral dynamics, pharmacology of available antiretroviral medications, and HIV-specific host responses. This is a Phase II trial to provide preliminary data on the feasibility and possible efficacy of using STI to enhance immune-based control of HIV-1 replication. A steady state HIV-1 viral load determined from historical tests prior to initiating highly active antiretroviral therapy (HAART) will be compared to the steady state viral load post-STI. HIV-1 specific CD4 and CD8 cell responses will be measured before and after the period of STI management and HIV-1 specific CD8 cell maturational phenotype will be assessed and correlated with ability to control viral replication.

Adolescents and young adults who have either had sustained viral suppression on HAART for at least 2 years or who have had sustained viral suppression from 3 to 6 months will be eligible for this study. Participants will have 12 weeks of HAART followed by 2 to 4 weeks of treatment interruption. Participants will undergo three rounds of this regimen. After the third STI, participants will have an additional 12 weeks of HAART and then stop therapy. Participants will be monitored off HAART for up to 20 weeks. During this time, if there is evidence of HIV progression (two consecutive viral loads exceeding 10,000 copies/ml; two consecutive CD4 cell counts under 350 cells/microL; two consecutive CD4 percentages less than 15%; or two consecutive CD4 cell counts less than 50% of baseline), standard continuous antiretroviral therapy will be reinstituted. Plasma HIV RNA will be tested monthly during therapy and weekly while subjects are off treatment. Immunologic studies are monthly throughout the study. Participants will be involved in the study for approximately 2 years.

ELIGIBILITY:
Inclusion Criteria

* Acquired HIV infection after age 12 years
* CD4 cell count greater than 500 cells/microL within 30 days of study entry
* Either on HAART for 3 to 6 months with HIV-1 RNA < 400 copies/ml or on HAART for more than 2 years with at least one HIV-1 RNA < 400 copies/ml each six month period
* HAART regimen of two NRTIs and at least one PI (not nelfinavir)
* HIV-1 RNA 5,000 copies/ml prior to HAART and documented CD4 cell values
* CMV positive
* Ability and willingness of subject (and parent/guardian where required) to give informed consent

Exclusion Criteria

* Started initial HAART regimen less than one year after known HIV-1 seroconversion
* Immunosuppressive therapy
* Certain medications
* Pregnancy
* Evidence of an opportunistic infection
* Laboratory values that are classified as Grade 3 or higher toxicities at the time of study enrollment

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2003-07

CONTACTS AND LOCATIONS:
Overall Officials: Craig M Wilson, MD, Study Chair — University of Alabama at Birmingham
Locations (4):
- United States (4):
  - University of California at San Diego, San Diego, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Diagnostic and Treatment Center, Fort Lauderdale, Florida
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- See also: Description of Adolescent Trials Networks (ATN) and contact information — http://www.atnonline.org